CLINICAL TRIAL: NCT06523569
Title: Mobile Health Interventions to Prevent Heart Disease After Hypertensive Disorders of Pregnancy
Acronym: mHEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Friends of Prentice (Other); Senior Faculty Academy (Unknown)
Responsible Party: Principal Investigator, Priya Freaney, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00219095
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hypertension in Pregnancy; Pre-Eclampsia; Eclampsia; Gestational Hypertension
Keywords: digital health; echocardiogram; blood pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Control) (No Intervention): Participant will receive usual care.
- Bundled digital health intervention (Experimental): Participant will be enrolled in a digital blood pressure monitoring program and receive a subscription to a mobile health lifestyle change application (Noom) alongside usual care.
  Interventions: Other: Digital Blood Pressure Monitoring System; Other: Mobile health application

INTERVENTIONS:
Other: Digital Blood Pressure Monitoring System — As a part of the bundled digital health intervention, the participant will receive instructions on how to follow a link in their electronic patient portal that will allow direct input of home blood pressure readings for clinical review.
  Arms: Bundled digital health intervention
Other: Mobile health application — As a part of the bundled digital health intervention, the participant will be given a lifestyle change mobile health application.
  Arms: Bundled digital health intervention

SUMMARY:
The purpose of this research is to study digital health interventions to prevent cardiovascular disease in individuals who have had a hypertensive disorder of pregnancy (HDP).

DETAILED DESCRIPTION:
The purpose of this research is to test the effect of two digital health interventions on cardiovascular health and subclinical cardiac dysfunction in postpartum individuals after pregnancies complicated by new-onset hypertensive disorder of pregnancy (HDP). All participants will undergo echocardiography and have their blood pressure/weight captured at 3 months and 12 months postpartum. If randomized to the intervention arm, the participant will be given a subscription to a mobile health application and a digital blood pressure monitoring system, and asked to utilize these at home during the one year of the study along with usual care. If randomized to the control arm, the participant will receive care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at Northwestern Memorial Hospital (Prentice Women's Hospital)
* Live birth at any gestational age
* Pregnancy complicated by new-onset HDP (pre-eclampsia, eclampsia, or gestational hypertension)

Exclusion Criteria:

* HELLP syndrome
* History of chronic diseases pre-pregnancy (hypertension, diabetes, cardiovascular disease, chronic renal disease)
* Current Omron remote patient monitoring or Noom user
* BMI<18.5 kg/m2 at enrollment
* Inadequate gestational weight gain or gestational weight loss

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 months postpartum; 12 months postpartum
  All participants will have systolic blood pressure measured at 3 months and 12 months postpartum

SECONDARY OUTCOMES:
Weight | 3 months postpartum; 12 months postpartum
  All participants will have weight measured at 3 months and 12 months postpartum
Subclinical cardiovascular dysfunction via echocardiography | 3 months postpartum; 12 months postpartum
  All participants will have echocardiography performed at 3 months and 12 months postpartum to assess subclinical cardiovascular dysfunction
Study feasibility | 12 months postpartum
  The investigators will assess study feasibility (% enrolled in digital health intervention) at the end of the study
Participant engagement | 12 months postpartum
  The investigators will assess participant engagement (% continuing to actively use digital health interventions) at the end of the study
Anti-hypertensive medication use (%) | 3 months postpartum; 12 months postpartum
  The investigators will assess participant anti-hypertensive medication use (%) at 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Priya M Freaney, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Dept. of Cardiology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No